CLINICAL TRIAL: NCT06633809
Title: Therapy Evaluation in Patients With Minor Stroke and Large Vessel Occlusion: A Prospective Multicenter Registry Study
Brief Title: Therapy Evaluation in Patients With Minor Stroke and Large Vessel Occlusion
Acronym: TEMPOS
Status: Recruiting | Type: Observational
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Jinhua Zhang, Prof., Sir Run Run Shaw Hospital
Other Study IDs: 20210607-34
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Stroke, Acute; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Vascular Diseases; Brain Infarction; Nervous System Diseases
Keywords: stroke; Mechanical thrombectomy; Proximal intracranial arterial occlusions; Large vessel occlusion; acute neurological deterioration; Outcome
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Vascular Diseases; Brain Infarction; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immediate Endovascular Therapy: The immediate endovascular therapy is performed immediately after stroke onset with any thrombectomy device usually used.
  Interventions: Other: Immediate endovascular therapy
- Best Medical Therapy: The best medical therapy is standard medical therapy, including intravenous fibrinolysis, anticoagulants or antiplatelet, but NOT including any endovascular therapies. The rescue endovascular therapies may be performed in case of acute neurological deterioration.

INTERVENTIONS:
Other: Immediate endovascular therapy — The best medical therapy includes intravenous fibrinolysis, anticoagulants or antiplatelet, but NOT any immediate endovascular therapies.
  Other Names: Best medical therapy
  Groups: Immediate Endovascular Therapy

SUMMARY:
This multicenter registry study, which record the therapy strategy and follows up these acute ischemic stroke (AIS) patients with low NIHSS and large vessel occlusion (LVO), is intended to provide the important data for therapy evaluation and prognostic prediction of the LVO patients with low NIHSS.

DETAILED DESCRIPTION:
It was reported that about two third of the stoke patients might present with minor or mild stroke symptoms. 20-40% of those minor stroke patients had large vessel occlusion (LVO). AIS patients with LVO and low NIHSS are common and has been associated with early neurological deterioration and worse outcomes. Until now, the best therapy strategy for the acute stoke patients with minor stroke and large vessel occlusion is unknown. Thus, we sought to (1) explore the potential predictors of acute neurological deterioration and 90-day clinical outcome; (2) and evaluate the best therapy strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Acute ischemic stroke patients of NIHSS 0-5 with 24 hours after onset
3. Proximal intracranial artery occlusion on NCCT/CTA or MRI/MRA showing occlusion of the intracranial ICA, M1, or proximal M2 vessel
4. Baseline ASPECTS ≥6 or infarct Core Volume of < 70 on NCCT/DWI/CTP
5. Pre-mRS≤1

Exclusion Criteria:

1. Any sign of intracranial hemorrhage on baseline CT/MR;
2. Seizures at stroke onset
3. Baseline blood glucose of <2.78 mmol or >22.20 mmol, or platelet count < 100,000/uL or serum creatinine levels > 3.0 mg/dL
4. Participation in any investigational study in the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke patients with minor stroke (NIHSS 0-5) and large artery occlusion.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale at 90 days | 90 days
  modified Rankin Scale at 90 days
acute neurological deterioration | 24 hours
  It is neurological deterioration of presumed ischemic origin with an NIHSS score increase of 4 points or more within the 24 hours after onset.

SECONDARY OUTCOMES:
Incidence of symptomatic intracerebral hemorrhage | 2-3 days
  Incidence of symptomatic intracerebral hemorrhage according to ECASS II criteria
patients with good outcome comparing the two treatment groups | 90 days
  Good outcome is defined as a score of 0-2 on the 90-day mRS

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided